CLINICAL TRIAL: NCT06481969
Title: Application of Autologous Adipose Stromal Vascular Fraction in the Treatment of Premature Ovarian Insufficiency
Acronym: aSVF-POI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rui Yang (Other)
Responsible Party: Sponsor-Investigator, Rui Yang, Clinical associate professor, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF2024-2-40911
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Female fertility; Premature Ovarian Insufficiency; Adipose stromal vascular fraction
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized to two groups at a ratio of 1:1- SVF protocol, and conventional protocol.
Who Masked: Outcomes Assessor
Masking Description: Due to the particularity of the treatment plan, the evaluator, namely the follow-up personnel who collect the postoperative medical history and the ultrasound evaluator, will be blinded in this trial to hide the grouping results. Blinding of participants and researchers is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A-SVF group (Experimental): Qualified participants will be randomized into either of two groups. Participants in this group will undergo lower abdominal liposuction, preparation of SVF and ovarian injection, other standard assisted reproductive treatments are similar and parallel between two groups.
  Interventions: Procedure: Lower abdominal liposuction and preparation of SVF; Procedure: Ovarian injection
- Group B-Control group (Other): Qualified participants will be randomized into either of two groups. Participants in this group will be treated according to the current clinical routine of the reproductive center, other standard assisted reproductive treatments are similar and parallel between two groups.
  Interventions: Procedure: Conventional IVF

INTERVENTIONS:
Procedure: Conventional IVF — Conventional In Vitro Fertilization (IVF) procedure and standard assisted reproductive treatments.
  Arms: Group B-Control group
Procedure: Lower abdominal liposuction and preparation of SVF — After lower abdominal liposuction (the liposuction volume is about 100 ml), the preparation and quality inspection of SVF will be completed by a laboratory with good manufacturing practice-approved facilities immediately. The adipose tissue will be cut into pieces of about 1mm3, and the equal volume of 0.1% collagenase I will be added to digest the adipose tissue. The digestion will be terminated after 40 minutes, followed by isolation, filtration, centrifugation, resuspension and dilution to obtain the SVF suspension. The test items, including bacteria, fungi, viruses and endotoxin, will be tested, and the expression of SVF surface markers, including CD45, CD34, CD31, CD11b, CD44, CD73, CD105 and CD90, will be detected by flow cytometry to ensure the quality of the SVF suspension. After about 4 hours of quality control and detection, the SVF suspension will be transported to the operating room on ice in a sealed incubator.
  Arms: Group A-SVF group
Procedure: Ovarian injection — Under ultrasound guidance, the SVF suspension will be injected into patients' bilateral ovaries. SVF with a total amount of (1~2)×107 cells from autologous fat tissue will be transplanted into each side of ovary. There are 3 injection points on each side of ovary, and 330±10μl SVF suspension will be administered at each point. The administration volume of each ovary will be 1ml in total. After injection, the patients will be required to lie flat for 2 hours to observe whether there would be adverse events.
  Arms: Group A-SVF group

SUMMARY:
A single-center, prospective, randomised controlled clinical trial (1:1 treatment ratio), designed to investigate the efficacy and safety of autologous SVF in improving the pregnancy outcome of infertile patients with POI.

DETAILED DESCRIPTION:
A single-center, large-scale, prospective, randomized controlled clinical trial will enroll 260 patients diagnosed with POI based on the inclusion and exclusion criteria from Peking University Third Hospital. Eligible participants will be randomized to two groups at a ratio of 1:1- SVF protocol, and conventional protocol.The participation in this study will be approximately 2 years with a total of 6 visits and 3 follow-up phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥20 and ≤39 years who have childbearing requirements.
* Cessation of menstruation or oligomenorrhea for at least 4 months
* Serum level of basal follicle stimulating hormone (FSH) >25 U/L at least 2 times (during the second to fourth day of the menstrual cycle or during amenorrhea; The interval between the two tests is 4 weeks)
* Serum level of Anti-Mullerian hormone (AMH) ≤1.1 ng/ml
* Women with intact uterus and bilateral adnexa.
* Voluntary participation and informed consent obtained.

Exclusion Criteria:

* Women with autoimmune diseases.
* Women with abnormal and uncontrolled thyroid function.
* Women with tumors in bilateral adnexa that are not clearly benign or malignant.
* Women with a history of malignant tumors, radiation therapy or chemotherapy.
* Women with a history of venous thrombosis or pulmonary embolism during the screening period.
* Women with severe illnesses that are not suitable for pregnancy, such as diseases of the circulatory system, urinary system, digestive system, endocrine system, respiratory system, immune system, mental or neurological system, etc.
* Women who continuously used systemic glucocorticoids or other immunosuppressants for≥3 weeks within 6 months before administration and women who used systemic glucocorticoids (prednisone≥20 mg/d or equivalent dose) or other immunosuppressants within 3 days before administration.
* Women who are allergic to the active ingredients or excipients of test drugs.
* Women with a family history of severe genetic diseases or gynecologic malignancies.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative clinical pregnancy rate in half a year | half a year after treatment
  Percentage of patients with clinical pregnancy within half a year after treatment

SECONDARY OUTCOMES:
Serum level of Anti-Mullerian hormone (AMH) | half a year after treatment
  Efficacy rate (%) = The number of patients with two consecutive increases in serum level of AMH after treatment / total number of included patients×100%
Antral follicles count (AFC) | half a year after treatment
  Efficacy rate (%) = The number of patients with bilateral ovarian AFC increases by at least 2 after treatment / total number of included patients×100%
Serum level of sex hormone (E2 and FSH) | half a year after treatment
  Efficacy rate (%) = The number of patients with two consecutive increases/decreases in serum level of E2/FSH after treatment / total number of included patients×100%
Ovarian volume | half a year after treatment
  Ovarian volume will be recorded before and after treatment. Paired sample t-test or independent sample t-test will be used to compare the changes in ovarian volume between the control and SVF treatment groups, P < 0.05 will be recorded as significant change in ovarian volume.
Menstrual status | half a year after treatment
  The frequency, duration and volume of menses within half a year after treatment will be recorded to evaluate whether the menstrual status of patients have improved. Menstrual recovery rate (%) = The number of patients with menstrual recovery after treatment / total number of included patients × 100%.
Pregnancy outcome | 2 years after treatment
  Live births or miscarriage of patients with successful pregnancy within half a year will be followed up. Live birth defined as the delivery of at least one viable fetus after 24 weeks gestation. Miscarriage defined as a loss of pregnancy before 24 weeks gestation. Live birth rate (%) = The number of patients with live births after treatment / total number of included patients×100%. Miscarriage rate (%) = The number of patients with miscarriage after treatment / total number of included patients×100%.
Health status of offspring | 2 years after treatment
  The health status (survival, physiological and intellectual development) of offspring will be followed up via telephone for 2 years.
Adverse reactions | 2 years after treatment
  The frequency, date of onset, duration and severity of any local and systemic adverse reactions will be observed and recorded during the entire follow-up period. Incidence rate of adverse reactions (%) = The number of patients with adverse reactions after treatment / total number of included patients×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Yang, M.D., Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Liu H, Lou Y, Li J, Liu C, Zhang H, Zhang C, Guo Q, Liu X, Yang W, Li J, Tian T, Zeng L, Xu H, Yang S, Zhen X, Bi H, Yang R, Yu Y, Ma C, Li R, Liu P, Qiao J. Efficacy and safety of autologous adipose tissue-derived stromal vascular fraction in patients with premature ovarian insufficiency: protocol for a single-centre randomised controlled trial. BMJ Open. 2025 Apr 3;15(4):e093804. doi: 10.1136/bmjopen-2024-093804. PMID 40180397